CLINICAL TRIAL: NCT04768465
Title: Effectiveness and Safety of Tacrolimus Combined With Low-dose Prednisone for Treatment of Myasthenia Gravis: A Real-world Study
Brief Title: Tacrolimus Combined With Low-dose Prednisone for Treatment of Myasthenia Gravis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Da, Yuwei, M.D. (Individual)
Responsible Party: Sponsor
Other Study IDs: 1.0
Record Dates: First submitted 2021-02-21; First posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Myasthenia Gravis
Keywords: myasthenia gravis; treatment; tacrolimus; low-dose prednisone
MeSH Terms: conditions — Myasthenia Gravis | interventions — Pyridostigmine Bromide; Prednisone; Tacrolimus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Blood samples are collected at baseline and 1, 3, 6 months after treatment initiation to monitor side effect and serum IL-2 level.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Combined Immunotherapy: MG patients are treated with tacrolimus combined with low-dose prednisone (0.25mg/kg/d).
  Symptomatic treatment like pyridostigmine bromide can be added to relieve symptoms (≤480mg/d).
  Interventions: Drug: Pyridostigmine, Prednisone, Tacrolimus
- Tacrolimus monotherapy: MG patients are treated with tacrolimus as initial immune monotherapy. Symptomatic treatment like pyridostigmine bromide can be added to relieve symptoms (≤480mg/d).
  Interventions: Drug: Pyridostigmine, Tacrolimus

INTERVENTIONS:
Drug: Pyridostigmine, Prednisone, Tacrolimus — Dose of tacrolimus should be initiated based on CYP3A5*3 polymorphism and adjusted to achieve blood trough concentration of 4.8-10.0 ng/ml. Prednisone is administrated with an initial dose of 0.25mg/kg/d and started to tamper with the achievement of MMS or the presence of any intolerable side effects. The rate of tampering is considered by the physician, usually no more than 5mg/month. If the participants failed to maintain MMS, dose of prednisone should be increased 5mg/week to 0.25mg/kg/d and maintained until MMS reached again. After MMS sustained for 1 month, prednisone dose would be tapered again with 2.5mg/month. Calcium and potassium supplements and gastric mucosa protectors could be addressed to avoid any adverse effects of prednisone. Treatment regimens are determined based on the physician's judgment and preferences of the patients. This study was observational and do not change the clinical course of patients.
  Other Names: Pyridostigmine Bromide; Deltacortone/Meticorten/Prednisone Acetate Tablets; Prograf/FK506
  Groups: Combined Immunotherapy
Drug: Pyridostigmine, Tacrolimus — Dose of tacrolimus should be initiated based on CYP3A5*3 polymorphism and adjusted to achieve blood trough concentration of 4.8-10.0 ng/ml. Treatment regimens are determined based on the physician's judgment and preferences of the patients. This study was observational and do not change the clinical course of patients.
  Other Names: Pyridostigmine Bromide; Prograf/FK506
  Groups: Tacrolimus monotherapy

SUMMARY:
This study is designed to evaluate the effectiveness and safety of tacrolimus combined with low-dose prednisone in the management of myasthenia gravis patients, compared to tacrolimus as initial immune monotherapy.

DETAILED DESCRIPTION:
This is a single center, observational real-world study recruiting myasthenia gravis patients from Neurology Departments of Xuanwu Hospital, aiming to compare effectiveness and safety of 2 different inmunotherapy for MG. The study plans to recruit 160 MG participants and divides into 2 treatment groups according to physician's judgment and preferences of patients, one is combined immunotherapy group in which tacrolimus added with low-dose prednisone (0.25mg/kg/d), and the other is tacrolimus monotherapy group. Both groups can be treated with pyridostigmine to relieve symptoms. Patients are followed up at 1, 3 and 6 month after treatment initiation to assess the efficacy of both regimen. The primary outcome is the change of MG-ADL scores. Also, liver and renal functions are tested to monitor any side effects. Patients' clinical records are uploaded to an online database.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Clinical Diagnosis of MG is confirmed based on typical clinical features of fluctuating muscle weakness, with at least 1 of the following supporting evidence:

  1. positive clinical response to acetylcholinesterase inhibitor
  2. positive AchR-Ab or MuSK-Ab testing
  3. decrement >10% in repetitive nerve stimulations study (RNS) or increased jitter on single-fibre electromyography (SFEMG)
* MGFA clinical classification: I - IV
* Baseline MG-ADL ≥ 3
* Disease course from onset to enrollment ≤ 12 months
* Cooperation to followup
* Written informed consent

Exclusion Criteria:

* Initiation of immunosuppressant for MG prior to screening, including Prednisone, Methylprednisolone, Azathioprine, Methotrexate, Cyclosporine A, Mycophenolate Mofetil, Tacrolimus and Cyclophosphamide
* Treatment of immunosuppressant for other concomitant disease 6 months prior to recruitment
* Rapid immunosuppressive treatments like Intravenous immunoglobulin or plasma exchange 1 month prior to recruitment
* Thymectomy within 3 months prior to Screening
* Concomitant chronic degenerative, psychiatric, or neurologic disorder that can cause weakness or fatigue
* Consciousness, dementia or schizophrenia
* Pregnancy or lactation, unwillingness to avoid pregnancy
* Uncontrolled hypertension or diabetes, Liver or kidney dysfunction, Cataract, Severe osteoporosis, Femoral head necrosis; Hyperkalemia, HIV, Acute or chronic infection
* Other conditions that would preclude participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Myasthenia Gravis
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Change of MG-specific Activities of Daily Living scale (MG-ADL) from Baseline | Baseline, 1 month, 3 months, 6 months
  The MG-ADL is an 8-item scale to assess symptoms of myasthenia gravis patients obtained by summing the responses to each individual item (Grades: 0,1,2,3). The score ranges from 0 to 24.

SECONDARY OUTCOMES:
Time to achievement of minimal manifestations (MMS) or better | From Baseline to 6 months
  The time duration from treatment initiation to the achievement of MMS or better. Clinical statuses of patients are assessed and categorized according to Myasthenia Gravis Foundation of America (MGFA) post-intervention status (PIS). MM or better includes Minimal Manifestation (MM), Pharmacologic Remission (PR) or Complete Remission (CR).
Time to achievement of Patient-Acceptable Symptom States | From Baseline to 6 months
  The Patient-Acceptable Symptom States question is a simple yes or no query that asked: "Considering all the ways you are affected by Myasthenia, if you had to stay in your current state for the next month, would you say that your current disease state status is satisfactory?" This question reflects the patients assessment of their own health.
Change of Quantitative Myasthenia Gravis (QMG) Scores from Baseline | Baseline, 1 month, 3 months, 6 months
  The QMG is a 13-item scale which measures ocular, bulbar, limb function and respiratory function. The total score ranges from 0 (no myasthenic findings) to 39 (maximal myasthenic deficits) obtained by summing the responses to each individual item (None=0, Mild=1, Moderate=2, Severe=3).
Change of Myasthenia Gravis Quantity-of-Life Scale (MG-QoL15) from Baseline | Baseline, 1 month, 3 months, 6 months
  The MG-QOL15 is helpful in informing the clinician about the patient's perception of the extent of and dissatisfaction with myasthenia gravis (MG)-related dysfunction. MG-QOL15 evaluates patients' aspects about physical status, social adaptation and mental well-being.
Changes of MG-ADL subscores from baseline | Baseline, 1 month, 3 months, 6 months
  Subscores of ADL items can reflect patients' assessment about different MG-related dysfunctions, including ptosis, diplopia, talking, chewing, swallowing, breathing and limbs function.
Serum IL-2 level | Baseline, 1 month, 3 months, 6 months
  Tacrolimus exerts its immunosuppressive effect by inhibiting the early phase gene expression during T-cell activation, including the pro-inflammation IL-2 gene. Thus serum IL-2 is tested as a target of tacrolimus and also a marker of in vivo auto-immune status after treatment.
Treatment Failure | Baseline to 6 months
  Treatment failure is defined as discontinuation of tacrolimus therapy in patients who failed to achieve MMS or better or suffered from exacerbations (MG-ADL or QMG scores increase 50%) or myasthenia crisis.
Withdrawal | Baseline to 6 months
  Participants quit the clinical trial for any reason including unsatisfied response, economic burden or poor compliance to treatment protocol. Patients may quit at any time they want.

CONTACTS AND LOCATIONS:
Overall Officials: Yuwei Da, M.D., Study Chair — Xuanwu Hospital, Beijing
Locations (1):
- Yuwei Da, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided